CLINICAL TRIAL: NCT03706716
Title: Support Women's Decision Making - the Effect of Using an Online App in the Clinical Consultations of Patients With Urogenital Prolapse. A Protocol for a Randomized Controlled Non Blinded Multicenter Study. Assessing Feasibility.
Brief Title: Testing a Decision Aid for Women With Urogenital Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: OP_613
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-04

CONDITIONS: Pelvic Organ Prolapse
Keywords: shared decision making
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: Arm A - intervention /consultation with use of decision aid Arm B - Controls / consultation without use of decision aid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention with use of decision aid in the consultation (Other): With use of developed decision aid for pelvic organ prolapse / At the beginning of the consultation the IF will be opened within the patients electronic journal. The conversation will take its starting point from the generated IF which should define the area of interest rather for the patient.
  Interventions: Other: decision aid developed for pelvic organ prolapse
- Control with no use of decision aid in the consultation (No Intervention): Without decision aid / The conversation during the consultation will follow the general standard for consultation conversations in the department.

INTERVENTIONS:
Other: decision aid developed for pelvic organ prolapse — Conversation based upon the inter face in the Electronic patient journal.
  Arms: Intervention with use of decision aid in the consultation

SUMMARY:
Development of a decision aid for women with urogenital prolapse followed by an intervention with use of the decision aid to investigate the effect on the perceived shared decision making in the clinical consultations.

A protocol for a randomized controlled non blinded multicenter trial. A feasibility trial for the protocol.

DETAILED DESCRIPTION:
Objective :

The objective is to develop a decision aid to increase successful patient involvement and increased health care professionals integration of preferences in the clinical consultations with women with urogenital prolapse.

Method:

in the context of consultations an online app solution using a multicriterial analytic approach is developed and tested in order to support shared decision making (SDM). The decision aid is developed involving four national gynecological departments through participatory design. The decision aid is tested in a randomized, controlled multicenter trial in three hospital departments in the Region of Southern Denmark. A feasibility trial for the protocol of a randomized controlled trial will decide for further approach in relations to testing the online app. in a larger scale In the randomized trial patients will either receive consultations as usual (controls) or consultations using the interface (IF) in an app. The IF is generated upon data from a patient survey regarding their preferences for treatment beforehand.

Effect measures are the perceived shared decision making within the consultation (SDM-Q-9 ) and the patientperceived satisfaction with the decision (SWD)

ELIGIBILITY:
Inclusion Criteria:

* urogenital prolaps symptoms
* e boks

Exclusion Criteria:

* complicated pelvic organ prolapse which requires treatment other than dialogue, pessary, cystocele or rectocele surgery, physiotherapy or local hormones
* physical status classification system (ASA) score 3 or above
* not able to understand Danish without interpreter
* recurrent pelvic organ prolapse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
PROM of the shared decision making process | 1 hour immediately after the decision on treatment was taken
  Measurement of shared decision making for treatment of pelvic organ prolapse symptoms measured by questionnaire SDM-Q-9

SECONDARY OUTCOMES:
PROM of Satisfaction with decision | 1 hour immediately after the decision on treatment was taken
  Measurement of satisfaction with the decision for treatment of pelvic organ prolapse symptoms measured by questionnaire SWD

CONTACTS AND LOCATIONS:
Overall Officials: Mette Hulbaek, Ph.d. stud., Principal Investigator — Gynecology dep, Southern hospital of Jutland
Locations (3):
- Denmark (3):
  - Hospital of Southern Jutland, Aabenraa
  - Hospital of Lillebaelt, Kolding, Kolding
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hulbaek M, Primdahl J, Birkelund R, Al-Kozai SAH, Barawi S, Ebbesen NT, Nielsen JB. A Preference-Sensitive Online Instrument to Support Shared Decision Making for Patients With Pelvic Organ Prolapse: A Pilot Multicenter Randomized Controlled Trial. Comput Inform Nurs. 2021 Jul 12;39(11):714-724. doi: 10.1097/CIN.0000000000000789. PMID 34238835